CLINICAL TRIAL: NCT04911114
Title: Targeted Physical Activity to Improve Mobility and Falls Risk in Women Living With Ovarian Cancer (The BE-BALANCED Study)
Brief Title: Targeted Physical Activity to Improve Mobility and Falls Risk in Women Living With Ovarian Cancer
Acronym: BE-BALANCED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Kristin Campbell, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H20-02654
Record Dates: First submitted 2021-03-22; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Ovarian Cancer
Keywords: Cancer; Supervised Exercise; Virtual; Healthy Eating
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective single-arm feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): This is a single arm pilot study of group base exercise
  Interventions: Behavioral: Be-Balanced

INTERVENTIONS:
Behavioral: Be-Balanced — The BE-BALANCED program will run for 12-weeks, with participants attending group-based virtual supervised exercise sessions twice weekly. Participants will complete an individual in-person assessment at baseline and again at end of intervention to collect physical outcome measures and will complete questionnaires electronically using REDCap, (or mailed version). Follow-up assessments will be administered electronically to each participant using REDCap at 3-months after program completion (24 weeks post-baseline).

SUMMARY:
This study will explore the feasibility (suitability), efficacy (research-setting outcomes), and participant satisfaction of a virtually-supervised 12-week exercise and diet intervention for women with ovarian cancer. It will include exercise, behavior change strategies, and guidance around healthy eating. Participants will be instructed and supervised virtually in two exercise sessions weekly for 12 weeks by a professional trained to deliver the program. An additional 1 exercise session per week, completed independently, will be added from weeks 4-12 of the program. Finally participants will participate in two separate virtual group nutrition sessions. Assessments will occur at baseline, end-of-intervention, and 6 months post-baseline.

DETAILED DESCRIPTION:
Purpose: To assess the feasibility, preliminary efficacy, and patient perspectives of a 12-week supervised, virtually-delivered exercise and healthy eating program for women living with and beyond ovarian cancer.

Hypothesis: The investigators hypothesize that the program will be feasible and will demonstrate efficacy, and that patient perspectives will be overall positive and in support of the program.

Justification: Women living with and beyond ovarian cancer exercise at levels below the general population, and are at an increased risk for falls. Exercise and healthy eating programming is not a part of routine care. This project has the potential to demonstrate a feasible and relatively low-cost option for offering such programming.

Objectives: the objectives of this program are: 1) Primary Objective: To measure the feasibility of delivering the BE-BALANCED program from a virtual (i.e. live video) setting. Feasibility will be evaluated per individual item based on a priori targets; 2) Secondary Objective: To evaluate the preliminary efficacy of the BE-BALANCED program; 3) Tertiary Objective: To evaluate patient satisfaction (post-intervention only)

Research Design: This study is a prospective single-arm feasibility study.

Statistical Analysis: The primary aim is feasibility. This will be evaluated using descriptive statistics, focusing on the program recruitment, attendance, attrition, and fidelity. For secondary and tertiary/exploratory aims, a repeated measures ANOVA will be performed for each measure to evaluate the change in outcomes from baseline and end of intervention (12-weeks) and 3-month follow-up. In addition to the RM-ANOVA, an effect size for each measure will be calculated based on the same time-frame comparisons. SPSS will be used to process data.

ELIGIBILITY:
Inclusion Criteria:

1. 50-75 years of age (women tend to be older at time of diagnosis, with a median age in Canada of 62 years);
2. Completed primary chemotherapy treatment (oral maintenance therapy allowed);
3. Are within one year of completion of primary chemotherapy without known recurrence;
4. Have access to a smartphone, tablet, laptop, or desktop computer with a camera and microphone, and a reliable internet connection;
5. Speak English, to ensure safety in delivery of the physical activity intervention

Exclusion Criteria:

1. Do not pass pre-exercise screening for safety and do not subsequently provide written medical clearance from their physician to participate;
2. Do not consent to adhere to safety requirements to participate in a virtual delivery program (i.e., be seen on video for duration of class);
3. Experienced a fall requiring medical attention in the prior 6 months as individuals may be a higher risk for fall in a virtual physical activity program setting and would be more appropriate for referral to falls clinic

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Accrual | Baseline (0 weeks)
  Assessed by meeting accrual targets (number recruited)
Intervention Adherence | Baseline to 12 weeks
  Assessed as number of supervised virtual sessions that a participant attended, out of a total of 24 group exercise sessions, and number of self-directed sessions completed, out of a total of 9 sessions.
Attrition | Baseline to 12 weeks
  Assessed as number of drop-outs during the 12-week program.
Fidelity of group belonging | Baseline to 12 weeks
  Group Belonging Scale (0-20; higher is better)

SECONDARY OUTCOMES:
Physical function: Gait speed | Change from baseline to 12 weeks (end of intervention)
  Measured by the gait speed portion of The Short Physical Performance Battery. Measured in seconds.
Physical function: Functional mobility | Change from baseline to 12 weeks (end of intervention)
  Measured by 8 foot timed up and go (Seniors Fitness Test). Measured by distance in seconds.
Physical function: Lower extremity strength and endurance | Change from baseline to 12 weeks (end of intervention)
  Measured by 30-second chair stand (Seniors Fitness Test). Measured in repetitions completed.
Physical function: Upper extremity strength and endurance | Change from baseline to 12 weeks (end of intervention)
  Measured by 30-second biceps curl (Seniors Fitness Test). Measured in repetitions completed.
Physical function: Balance | Change from baseline to 12 weeks (end of intervention)
  Measured by Functional Reach Test. Measured in centimeters.
Cardiovascular Fitness | Change from baseline to 12 weeks (end of intervention)
  Measured by the Six Minute Walk test. Measured in meters.
Height | Change from baseline to 12 weeks (end of intervention)
  Measured using stadiometer. Measured in meters
Weight | Change from baseline to 12 weeks (end of intervention)
  Measured using a scale. Measured in kilograms
Body mass index | Change from baseline to 12 weeks (end of intervention)
  Aggregated measure of height and weight, reported in kilograms/meter^2
Waist circumference | Change from baseline to 12 weeks (end of intervention)
  Measured in centimeters
Hip circumference | Change from baseline to 12 weeks (end of intervention)
  Measured in centimeters
Health-related quality of life: Physical Health | Change from baseline to 12 weeks (end of intervention)
  Measured by 36-item Short Form Health Survey; Norm-based 0-100, higher score represents better health
Health-related quality of life: Mental Health | Change from baseline to 12 weeks (end of intervention)
  Measured by 36-item Short Form Health Survey; Norm-based 0-100, higher score represents better health
Depression and anxiety | Change from baseline to 12 weeks (end of intervention)
  Measured by Hospital Anxiety and Depression Scale; Score range 0-21, higher score is higher depression and anxiety.
Usual physical activity levels | Change from baseline to 12 weeks (end of intervention)
  Measured by Modified Godin Leisure Time Physical Activity questionnaire; Scoring range 0 - no specified maximum. Scoring < 14 units "insufficiently Active" ; 14-23 is "moderately active" and >=24 is "active".
Falls | Change from baseline to 12 weeks (end of intervention)
  Measured by standard falls calendar for the duration of the study as number of falls.

OTHER OUTCOMES:
Evaluate patient satisfaction | Baseline to 12 weeks
  Overall satisfaction; measured on scale 0-7 with higher score meaning higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Campbell, Principal Investigator — Department of Physical Therapy
Locations (1):
- Clinical Exercise Physiology Lab, Vancouver, British Columbia, Canada